CLINICAL TRIAL: NCT06776939
Title: Physiological Effect High-flow Tracheal Oxygen on Viscosity of Airway Mucus and Respiratory Effort in Patients Weaning from Invasive Mechanical Ventilation
Acronym: PIONEER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henrik Endeman (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor-Investigator, Henrik Endeman, Intensivist, Assistant professor Intensive Care, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MEC-2024-0468; NL87502.078.24 (Other: ABR)
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Weaning from Mechanical Ventilation; Tracheostomy Weaning; Respiratory Failure
Keywords: weaning from mechanical ventilation; tracheostomy; high flow oxygen; airway mucus; respiratory effort; dyspnea
MeSH Terms: conditions — Respiratory Insufficiency; Dyspnea | interventions — Oxygen Inhalation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- First high-flow tracheal oxygen, then conventional oxygen therapy (Active Comparator): The disconnection sessions on the days with study measurements are started with high-flow tracheal oxygen, and the second disconnection session is supported with conventional oxygen therapy. Conventional oxygen therapy is provided using a heat-moisture exchanger.
  Interventions: Device: Oxygen therapy
- First conventional oxygen therapy, then high-flow tracheal oxygen (Active Comparator): The disconnection sessions on the days with study measurements are started with conventional oxygen therapy, and the second disconnection session is supported with high-flow tracheal oxygen. Conventional oxygen therapy is provided using a heat-moisture exchanger.
  Interventions: Device: Oxygen therapy

INTERVENTIONS:
Device: Oxygen therapy — All patients are subject to both oxygen therapy groups in this randomized cross-over study. Study measurements are performed during several different disconnection sessions. Disconnection sessions can either be short (<90 min) or long (12 hours). Both short and long disconnection sessions are performed twice; once with conventional oxygen, and once with high-flow tracheal oxygen as respiratory support.

SUMMARY:
Rationale: Tracheostomized patients weaning from mechanical ventilation are at risk for dryness of airway mucosa and sputum accumulation during disconnection from mechanical ventilation. High-flow tracheal oxygen (HFTO) is being used as supportive therapy during disconnection sessions in tracheostomized patients weaning from invasive mechanical ventilation (IMV) to limit dryness while maintaining oxygenation. We recently summarized the studies comparing physiological effects HFTO as compared to other interfaces, collectively referred to as conventional oxygen therapy (COT), in a systematic review and identified areas of lacking knowledge: effect on sputum viscoelasticity, respiratory effort early in the weaning process and dyspnea sensation. We hypothesize that HFTO, compared to COT, decreases viscoelasticity of the sputum and provides respiratory support during weaning. This may improve weaning by facilitating clearance of airway mucus, preventing respiratory failure, and providing comfort by decreasing dyspnea.

Objective: To determine the physiological effect of HFTO compared to COT on sputum viscoelasticity, respiratory effort and dyspnoea.

Study design: Pilot study with randomized crossover design, single-center. Study population: Twenty adult patients weaning from mechanical ventilation with tracheostomy.

Intervention (if applicable): Crossover with COT and HFTO during two days in the weaning phase.

Main study parameters/endpoints: Primary endpoint: sputum viscoelasticity measured by rheology during long disconnection sessions in the final phase of weaning. Secondary endpoints: respiratory effect measured by swings in esophageal pressure (PES) and prevalence and severity of dyspnoea sensation by visual analogue scale (VAS).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The study compares two therapeutic modalities both used in clinical care without side-effects or complications. Study procedures and measurements consist of standard clinical procedures that are performed daily in clinical setting with negligible risk of deterioration for the patient. During weaning with HFTO sputum clearance might be more easy for the patient and respiratory effort might decrease, both are assumed to be beneficial for the weaning process of the patient.

ELIGIBILITY:
Inclusion:

* Age ≥18 years
* Weaning from mechanical ventilation with tracheostomy

Exclusion Criteria:

* Longstanding tracheostomy, defined as tracheostomy being present prior to current hospital admission
* Tracheostomy primarily indicated for chronic upper airway obstruction or to secure airway patency due to persistent stupor/coma
* Chronic positive pressure respiratory support at home (excluding night-time continuous positive airway pressure for sleep apnea)
* Mucociliary disease in medical history (e.g. cystic fibrosis, pulmonary ciliary dyskinesia)
* Neuromuscular disease in medical history (excluding ICU-acquired weakness)
* Contra-indication placement oesophageal balloon for measurement of PES, such as:

  * Fractures in mandibular, orbital or ethmoid bone or skull base
  * Esophageal varices or surgery in medical history
  * Severe bleeding disorders
* Hemoptysis in 72 hours prior to the first disconnection session. Clinically relevant hemoptysis is defined as hemoptysis requiring tracheal/endobronchial or radiologic intervention, or administration of pro-coagulating drugs such as tranexamic acid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Sputum viscoelasticity | The 12-hour disconnection session
  During disconnection from the ventilator patients do not breathe actively heated and humidified gas mixtures. During disconnection from the ventilator the airway mucus thickens. This thickening can be quantified by measuring visco-elasticity and at the end of the disconnection sessions. The change in visco-elasticity between the start and end of the disconnection session will be compared within patients between disconnection sessions with HME and HFTO. Hence, the primary end-point is the change in sputum viscoelasticity from baseline to the end of the long disconnection sessions (≥12 hours). Viscoelastic (G*) is made up of elasticity (G') and viscosity (G'') of mucus at a 5% strain rate (or linear viscoelastic region, which reflects the small deformation regime) and the critical stress (σ critical)· and strain (y critical) of mucus, which reflect the behavior of mucus under high amounts of shear stress and thus the large deformation regime.

SECONDARY OUTCOMES:
Sputum visco-elasiticity | The short disconnection session (<90 minutes)
  The difference between COT and HFTO in change in sputum viscoelasticity from baseline to the end (after 10-90 min) of the early disconnection session
Dyspnea presence | At early (<90 min) and late (12 hour) disconnection sessions
  The presence of self-reported dyspnea sensation during early (<90 min) and late (12 hour) disconnection sessions. Presence of self-reported dyspnea and discomfort is evaluated by asking patients.
Respiratory effort | The short disconnection session (<90 minutes)
  The difference in respiratory effort between conventional oxygen therapy and high-flow oxygen therapy during early disconnection sessions measured by median esophageal pressure swing and pressure time product during the early disconnection session.
Dyspnea severity | early (<90 min) and late (12 hour) disconnection sessions
  The severity of self-reported dyspnea sensation during early (<90 min) and late (12 hour) disconnection sessions. Severity of self-reported dyspnea is evaluated using a dyspnea visual-analog scale (D-VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided